CLINICAL TRIAL: NCT00783523
Title: Influence of Matrix Metalloproteinase on Brain Arteriovenous Malformation Hemorrhage
Brief Title: Influence of MMP on Brain AVM Hemorrhage
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: H42145-30334-02; AHA #0730360N
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Arteriovenous Malformations; Cavernous Angiomas; Brain Aneurysms
MeSH Terms: conditions — Arteriovenous Malformations; Hemangioma, Cavernous; Intracranial Aneurysm | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doxycycline (Active Comparator): Patients undergoing elective vascular malformation surgery will receive doxycycline100 mg twice a day, a dose shown to effectively decrease MMP or placebo, treatment for two weeks prior to surgery
  Interventions: Drug: Doxycycline or Placebo
- Placebo (Placebo Comparator): Patients undergoing elective vascular malformation surgery will receive doxycycline100 mg twice a day, a dose shown to effectively decrease MMP or placebo, treatment for two weeks prior to surgery
  Interventions: Drug: Doxycycline or Placebo

INTERVENTIONS:
Drug: Doxycycline or Placebo — Randomized to Doxycycline 100mg 2x/day or Placebo 2x/day for 1 or2-weeks pre-operatively.
  Other Names: Doxycycline; Placebo

SUMMARY:
Brain vascular malformations, including arteriovenous malformations (AVM), cavernous malformations (CVM) and aneurysms, are a source of life-threatening risk of intracranial hemorrhage. The etiology and pathogenesis are unknown. There is no medical therapy presently available. Prevention of spontaneous intracerebral hemorrhage (ICH) is the primary reason to treat brain vascular malformations. The goal of this study is to: begin pilot studies to lay the groundwork for future clinical trials to develop medical therapy to decrease ICH risk.

Matrix metalloproteinases (MMPs) regulate the extracellular matrix in association with various hemorrhagic brain disorders. MMP-9 has been most consistently associated with vascular wall instability and hemorrhagic brain disorders. Doxycycline, a non-specific MMP inhibitor, may enhance vascular stability, thus reducing the risk of spontaneous hemorrhage in brain vascular malformations by decreasing MMP-9 activity.

DETAILED DESCRIPTION:
* Doses will be randomized by the Pharmacy Department at UCSF for Doxycycline 100 mg/BID and Placebo BID. These will be prepared in blister-packs.
* Depending on enrollment/surgery date, patients will take medication either one to two weeks before surgery. Patients will be assigned to a treatment group according to a random table.
* Each patient will be initially provided with a 1 or 2-week supply of drug in blister packs. The patient will take the final dose of study drug on the morning of surgery.

Baseline labs will be obtained and then again at time of surgery along with a piece of surgical tissue.

ELIGIBILITY:
Inclusion Criteria:

* 13 years or older
* Female patients of child bearing age using barrier-type birth control
* Creatinine no greater than 2.0 mg/di
* Alanine aminotransferase (ALT) no greater than 2 times upper limit of normal
* WBC count at least 3,800/mm3
* BMI within 50% of normal

Exclusion Criteria:

* Allergy to tetracycline
* Unstable medical illness (unstable angina, advanced cancer, etc) over the last 30 days
* Female patients of child-bearing age not using effective birth control (barrier)
* History of vestibular disease (except benign positional vertigo)
* History of noncompliance with treatment or other experimental protocols
* Patients taking other antibiotics
* History of systemic lupus erythematosis
* Patients who are immunocompromised Patients with clinically significant hepatic dysfunction

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Our primary aim is to perform a pilot study to document the effect of doxycycline therapy to decrease MMP expression in the vascular malformation tissue. | 1 to 2-week pre-operative

SECONDARY OUTCOMES:
Our secondary aims are: (1) To explore whether plasma MMP-9 levels can be used as a marker for MMP-9 inhibition in the vascular malformation lesional tissue | 1 to 2-week pre operative

CONTACTS AND LOCATIONS:
Overall Officials: Chanhung Lee, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States